CLINICAL TRIAL: NCT05247645
Title: Structured Collection of Data Relating to Rare Diseases With Predominantly Skeletal Involvement
Brief Title: Data Collection of Patients With Rare Bone Diseases
Acronym: RD-DATA
Status: Recruiting | Type: Observational
Sponsor: Luca Sangiorgi (Other)
Responsible Party: Sponsor-Investigator, Luca Sangiorgi, Head of Department of Rare Skeletal Disorders, Istituto Ortopedico Rizzoli
Organization: Istituto Ortopedico Rizzoli (Other)
Other Study IDs: 792/2020/Oss/IOR
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Skeletal Dysplasia
Keywords: Rare Disease with predominantly skeletal involvement; Disease Evolution; Data Collection; Natural History Study
MeSH Terms: conditions — Mucopolysaccharidosis IV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Whole peripheral blood, DNA, lymphocytes, saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rare diseases with predominantly skeletal involvement: The group comprises all patients affected by rare diseases with predominantly skeletal involvement

SUMMARY:
RD-DATA is a retrospective and prospective data collection, finalized for care and research purposes. It is articulated in main sections - strongly related and mutually dependent on each other - corresponding to different data domains: personal information, clinical data, genetic data, genealogical data, surgeries, etc.

This approach has been developed to corroborate and integrate data from different sources and evaluating several aspects of the diseases and to correlate genetic background and phenotypic outcomes, in order to better investigate diseases pathophysiology. Due to legal requirements, institutional directives and organizational issues, we are unable to include individuals residing outside Italy in the registry at this time. We are currently engaged in the preparation of a recruitment process for individuals residing outside Italy.

DETAILED DESCRIPTION:
The traditional method of collecting patient information is frequently chaotic, inconvenient and sometimes even unsafe, particularly when dealing with rare diseases. In 2020, the need to simplify the diagnostic process and to overcome the difficulties of data storage and analysis, led to the suggestion of implementing the Data Collection of Patients With Rare Bone Diseases - RD-DATA.

The RD-DATA relies on an IT platform named Genotype-phenotype Data Integration platform (GeDI).This solution, realized by a collaboration among Rare Skeletal Disorders Department and a local software-house (Dilaxia Spa) is a General Data Protection Regulation (GDPR)-compliant, multi-client, web-accessible system and it has been designed according to current medical informatics standards (Orphanet code, ICD-10 (International Disease Classification), Human Genome Variants Society). GeDI is continuously implemented to improve management of persons with rare conditions with predominantly skeletal involvement and to help researchers in analysing collected information. RD-DATA is articulated in main sections:

Personal data: it comprises general information, birth details and residence data; Patient data: including the patients internal code, the hospital code and other details on patients; Diagnostic Process: the diagnosis, the status (affected, suspected, etc.), age at diagnosis, comorbidities, allergies, etc.; Genogram: a tool for designing family transmission of the disease, alongside information on the diseases status of all relatives included.

Clinical events: it records a long list of signs and symptoms as well as several additional items to describe the disease Genetic Analysis and Alteration: including technique, sample information, analysis duration, etc. In addition, this section comprises detailed information on detected pathological variants (gene, international reference, DNA change, Protein change, genomic position, etc.).

Visits: it includes the typology of the visit (genetic, orthopedic, rehabilitation, pediatric, etc.), the date of the visit, treatment, prescription, imaging, etc.

Treatments: this section comprises information of a wide range of treatments including pharmacological, devices, supplements, and other treatments such as psychological, nutritional, etc.; Documents: this repository allow us to store all types of documents (radiological reports, imaging, consents, clinical reports, etc.); Consents: this section provides a comprehensive overview of all consents collected, including the collection date; Samples: this section includes information on the samples, like the type, date of collection, etc.; PROs: this section collects information on patients reported outcomes such as the quality of life or ABC scale.

ELIGIBILITY:
Inclusion Criteria:

* All patients affected by rare diseases with predominantly skeletal involvement

Exclusion Criteria:

* Any condition unrelated to rare diseases with predominantly skeletal involvement

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The population has been individuated as all the patients in charge to Rare Skeletal Disorders Department affected by rare diseases with predominantly skeletal involvement
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-10-10 (Actual); Primary Completion 2045-10-09 (Estimated); Study Completion 2045-10-09 (Estimated)

PRIMARY OUTCOMES:
Natural History and Epidemiology in terms of clinical, genetic and functional evaluation | Since the disease is rare, the timeframe is strictly related to patients enrolment and consequently to amount of collected data. A 10 years period will probably answer general issues.
  To maintain an established registry in order to assess epidemiology and natural history.
  Collection of:
  1. physical examinations data: assessment of severity of the disease
  2. orthopedic and functional data: stature (cm), weight (kg), number and localization of sites affected by signs and symptoms, definition of deformities (localization and number), definition of limitations (localization and number)
  3. surgical procedures: type, number and site of surgeries disease-related and age at surgeries
  4. genetics background: target gene, type of mutation, type of variant detected, clinical significance
  5. family history: inheritance in maternal or paternal line
  6. treatment information: pharmacological, devices, supplements, and other treatments
  Clinical, orthopedic and functional features are updated at each follow up. Clinical reports, medical charts and imaging are the primary sources of data.

SECONDARY OUTCOMES:
Genotype-Phenotype Correlation among clinical features and eventual molecular background | 25 years
  The secondary outcome comprises the correlation between genotype and phenotype. This includes but is not limited to clinical features and genetic background. This will be pursued using the information collected during visits and follow-ups and the genetic information resulting from molecular investigations, when available.

OTHER OUTCOMES:
Longitudinal study of disease evolution (including prospective and retrospective data) | 25 years
  This outcome aims to investigate the evolution of the diseases. Main clinical features, such as height (cm), number and localization of signs and symptoms, number and localization of deformities, number and localization of limitations will be collected both retrospectively and prospectively in the entire population via physical examination, clinical reports and imaging.
  An evaluation of these parameters will be performed at each visit to keep track on the progression of the clinical manifestations.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Sangiorgi, MD, PhD, Principal Investigator — IRCCS istituto Ortopedico Rizzoli
Locations (1):
- Irccs Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

REFERENCES:
- See also: Rare Skeletal Disorders Department website — https://www.ior.it/index.php/en/curarsi-al-rizzoli/rare-skeletal-disorders